CLINICAL TRIAL: NCT02971735
Title: Cognitive Style and Mobile Technology in E-learning in Undergraduate Medical Education- A Randomized Controlled Trial of Otolaryngology-head and Neck Surgery
Brief Title: Cognitive Style and Mobile Technology in E-learning in Undergraduate Medical Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 105-5290C
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2016-11

CONDITIONS: Medical Education
Keywords: cognitive style; e-learning; mobile technology; randomized controlled trial; otolaryngology-head and neck surgery

STUDY DESIGN:
Intervention Model Description: This study was a prospective randomized controlled trial.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interactive multimedia module (Experimental): Subjects allocated to this experimental group will receive an intervention of mobile technology of e-learning (M-TEL) using the interactive multimedia (IM) module consist of integrated text, images, and small game tests (intervention) for 100 minutes. The module is a non-linearity of learning with interaction (student-based choice and pop-up feedback). This context has been adjusted to the same level to that of the PPS module.
  Interventions: Other: mobile technology of e-learning (M-TEL)
- Power Point show module (Active Comparator): Subjects allocated to this experimental group will receive an intervention of mobile technology of e-learning (M-TEL) using the Power Point show (PPS) module consist of integrated text, images, and audio (intervention) for 100 minutes. The module is a linear learning without interaction. This context has been adjusted to the same level to that of the IM module.
  Interventions: Other: mobile technology of e-learning (M-TEL)

INTERVENTIONS:
Other: mobile technology of e-learning (M-TEL) — UME students learn the Top 10 emergent ORL-HNS disorders using the M-TEL including the IM module or the PPS module.

SUMMARY:
New designs of 6-year undergraduate medical education (UME) in Taiwan mainly include (1) integral curricula of body organ system, (2) multiple methods of clinical teaching and assessment, and (3) generalism in UME. Accompany with decreasing educational hours in the classrooms and hospital, essential but minor components of primary healthcare such as ophthalmology and otolaryngology-head and neck surgery (ORL-HNS) is disproportionately under-represented in UME. Novel medical education stresses on enabling self-directory learning and increasing learning hours outside the classrooms. Accordingly, we hypothesize that innovations in educational technology can enhance the learning outcomes of ORL-HNS. This study is aimed to determine whether mobile technology in e-learning (M-TEL) is an effective tool for the instruction of ORL-HNS and to compare effects of different cognitive styles on learning outcomes of M-TEL with various modules of medical education. This is a randomized controlled trial. We will recruit 60 UME students without previous training in ORL-HNS to undergo the Group Embedded Figures Test to determine their cognitive styles such as field dependence or field-independence. After blinded randomization, students are instructed on two modules of emergent ORL-HNS disorders, using either a standard e-learning of text-figure Power Point show or an interactive multimedia module. Subjects are evaluated on emergent ORL-HNS disorders using text-based assessment and multimedia assessment take place prior to and following instruction. After 7 days later, they will be assessed using global satisfaction score and AttrakDiff2 questionnaire. We anticipate that this study can confirm M-TEL can enhance the efficiency of the instruction of ORL-HNS and understand differences in learning outcomes of M-TEL with various modules of medical education between field dependence and filed independence using this platform.

DETAILED DESCRIPTION:
Background:

New designs of 6-year undergraduate medical education (UME) mainly include (1) integral curricula of body organ system, (2) multiple methods of clinical teaching and assessment, and (3) generalism in UME. UME is meant to enable graduates to become undifferentiated general physicians. Accompany with decreasing educational hours in the classrooms and hospital, essential but minor components of primary healthcare such as ophthalmology and otolaryngology-head and neck surgery (ORL-HNS) is disproportionately under-represented in UME. In Canada, substantial downstream effects on managing ORL-HNS problems have been noted in family medicine residents. In order to improve learning insufficiency and enhance clinical competency without increasing extra-hours in the classrooms and hospitals, novel medical education stresses on enabling self-directory learning and increasing learning hours outside the classrooms. Accordingly, we hypothesize that innovations in educational technology can enhance the learning outcomes of ORL-HNS.

Purposes: This study is aimed to determine whether mobile technology in e-learning (M-TEL) is an effective tool for the instruction of ORL-HNS and to compare effects of different cognitive styles on learning outcomes of M-TEL with various modules of medical education.

Material and Methods:

This is a randomized controlled trial. Firstly, we have been setup a e-learning platform of the Top 10 emergent ORL-HNS disorders with translating into an application (APP) function that can execute in mobile devices. Secondly, we will recruit 60 UME students without previous training in ORL-HNS to undergo the Group Embedded Figures Test to determine their cognitive styles such as field dependence or field-independence. After blinded randomization, students are instructed on two modules of emergent ORL-HNS disorders, using either a standard e-learning of text-figure Power Point show or an interactive multimedia module. Subjects are evaluated on emergent ORL-HNS disorders using a text-based assessment and a multimedia assessment take place prior to and following instruction.

Anticipating Outcome:

This study can (1) establish a M-TEL of ORL-HNS that can deliver an innovatively mobile e-learning to supplement the deficiency of the classroom hours, (2) confirm M-TEL can enhance the efficiency of the instruction of ORL-HNS, and (3) understand differences in learning outcomes of M-TEL with various modules of medical education between field dependence and filed independence using this platform.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20 years old;
2. UME students (defined as the three or four years of medical school training).

Exclusion Criteria:

1. Previous ORL-HNS training;
2. Declining to participate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-23; Primary Completion 2017-07-05 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ang Lee, M.D., Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No
The individua participant data of UME students may be not suitable to be available to other researchers

REFERENCES:
- [Background] Glicksman JT, Brandt MG, Parr J, Fung K. Needs assessment of undergraduate education in otolaryngology among family medicine residents. J Otolaryngol Head Neck Surg. 2008 Oct;37(5):668-75. PMID 19128674
- [Background] Wolff M, Wagner MJ, Poznanski S, Schiller J, Santen S. Not another boring lecture: engaging learners with active learning techniques. J Emerg Med. 2015 Jan;48(1):85-93. doi: 10.1016/j.jemermed.2014.09.010. Epub 2014 Oct 13. PMID 25440868
- [Background] Yavner SD, Pusic MV, Kalet AL, Song HS, Hopkins MA, Nick MW, Ellaway RH. Twelve tips for improving the effectiveness of web-based multimedia instruction for clinical learners. Med Teach. 2015 Mar;37(3):239-44. doi: 10.3109/0142159X.2014.933202. Epub 2014 Aug 11. PMID 25109353
- [Background] Alegria DA, Boscardin C, Poncelet A, Mayfield C, Wamsley M. Using tablets to support self-regulated learning in a longitudinal integrated clerkship. Med Educ Online. 2014 Mar 12;19:23638. doi: 10.3402/meo.v19.23638. eCollection 2014. PMID 24646438
- [Background] Chapman DM, Calhoun JG. Validation of learning style measures: implications for medical education practice. Med Educ. 2006 Jun;40(6):576-83. doi: 10.1111/j.1365-2929.2006.02476.x. PMID 16700774
- [Derived] Lee LA, Wang SL, Chao YP, Tsai MS, Hsin LJ, Kang CJ, Fu CH, Chao WC, Huang CG, Li HY, Chuang CK. Mobile Technology in E-Learning for Undergraduate Medical Education on Emergent Otorhinolaryngology-Head and Neck Surgery Disorders: Pilot Randomized Controlled Trial. JMIR Med Educ. 2018 Mar 8;4(1):e8. doi: 10.2196/mededu.9237. PMID 29519776
- [Derived] Lee LA, Chao YP, Huang CG, Fang JT, Wang SL, Chuang CK, Kang CJ, Hsin LJ, Lin WN, Fang TJ, Li HY. Cognitive Style and Mobile E-Learning in Emergent Otorhinolaryngology-Head and Neck Surgery Disorders for Millennial Undergraduate Medical Students: Randomized Controlled Trial. J Med Internet Res. 2018 Feb 13;20(2):e56. doi: 10.2196/jmir.8987. PMID 29439943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 consecutive volunteers were recruited from a teaching clinic for the validation study from November 23, 2016 to July 5, 2017.
Pre-assignment Details: All of the volunteers had at least a basic level of computer literacy, and they were shown the practical aspects of using tablets and applications. The inclusion criteria were as follows: 1) age >20 years; and 2) undergraduate medical students (clerkship). The exclusion criteria were: 1) previous ORL-HNS training; and 2) declining to participate.
Period: Overall Study
Arm/Group | Interactive Multimedia Module | Power Point Show Module
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pretests including a 15-minute 10-question standard MCQ to evaluate the students' existing knowledge (range, 0-100) and a 15-minute 5-question MST to assess their existing competence (range, 0-100) with regards to "emergent ORL-HNS disorders" were given to the students.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interactive Multimedia Module | Power Point Show Module | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [23 to 24] | 23 [23 to 24] | 23 [23 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 20 | 16 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
The cognitive style was assessed using the 25-item group embedded figures test after enrollment. [Median (Inter-Quartile Range); unit: units on a scale] — The cognitive style of the participants was assessed using the 25-item GEFT after enrollment. On the basis of the number of correct answers given by the participants, the GEFT scores ranged from 0 (the most field-dependent [FD]) to 18 (the most field-independent [FI]). We stratified the students into two subgroups: "classical FD" (GEFT score ≤12) and "classical FI" (GEFT score >12).
  units on a scale | 18 [15 to 18] | 17 [16 to 18] | 17 [15 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Multiple-choice Question (MCQ) Scores
Description: Subjects will undergo the duplicated 15-minute MCQ tests before after the M-TEL Subjects will undergo the duplicated 15-minute MCQ tests 15 minutes before the M-TEL intervention with either the IM module or the PPS module and immediately after the M-TEL intervention.
Time Frame: before and immediately after the M-TEL intervention
Measure: Median (Inter-Quartile Range); unit: percentage of MCQ change
Arm/Group | Interactive Multimedia Module | Power Point Show Module
Number analyzed (Participants) | 30 | 30
percentage of MCQ change | 40 [13 to 76] | 45 [30 to 50]

2. Secondary Outcome: Percentage Change in Multimedia Situation Test (MST) Scores
Description: Subjects will undergo the duplicated 15-minute MST tests 15 minutes before the M-TEL intervention with either the IM module or the PPS module and immediately after the M-TEL intervention.
Time Frame: before and immediately after the M-TEL intervention
Measure: Median (Inter-Quartile Range); unit: percentage of MST change
Arm/Group | Interactive Multimedia Module | Power Point Show Module
Number analyzed (Participants) | 30 | 30
percentage of MST change | 0 [-21 to 38] | 25 [0 to 33]

3. Secondary Outcome: Global Satisfaction Score
Description: Global satisfaction score is measured using a visual analogue scale from 0 (very dissatisfied) to 10 (very satisfied) after 7 days post M-TEL.
Time Frame: 7 days after the M-TEL intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interactive Multimedia Module | Power Point Show Module
Number analyzed (Participants) | 30 | 30
score on a scale | 8 [6 to 9] | 6 [4 to 7]

4. Secondary Outcome: AttrakDiff2 Questionnaire: Pragmatic Quality Score
Description: For more delicately evaluate the acceptance of technical innovations, we will assess "user experience" using the AttrakDiff2. AttrakDiff2 is developed as a tool by Hassenzahl's research group to be able to quantify attractive, identifiable, stimulating, and pragmatic qualities. The tool consists of 28 seven-step items whose poles are opposite adjectives (e.g. "confusing - clear", "unusual - ordinary", "good - bad"). Each set of adjective items is ordered into a scale of intensity. Each of the mean values of an item group creates a scale value for pragmatic quality (PQ), hedonic stimulation (HQ-S), hedonic identification (HQ-I), and attractiveness (ATT) (range: -3-3).
Time Frame: 7 days after the M-TEL intervention
Population: Pragmatic quality
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interactive Multimedia Module | Power Point Show Module
Number analyzed (Participants) | 30 | 30
score on a scale | 1.7 [0.7 to 2.3] | 0.0 [-0.6 to 1.3]

5. Secondary Outcome: AttrakDiff2 Questionnaire: Hedonic Stimulation
Description: as for outcome 4
Time Frame: 7 days after the M-TEL intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Interactive Multimedia Module | Power Point Show Module
Number analyzed (Participants) | 30 | 30
units on a scale | 1.5 [0.6 to 2.0] | -0.3 [-1.0 to 0.9]

6. Secondary Outcome: AttrakDiff2 Questionnaire: Hedonic Identification
Description: as for outcome 4
Time Frame: 7 days after the M-TEL intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Interactive Multimedia Module | Power Point Show Module
Number analyzed (Participants) | 30 | 30
units on a scale | 1.4 [0.7 to 2.0] | 0.3 [-0.2 to 1.2]

7. Secondary Outcome: AttrakDiff2 Questionnaire: Attractiveness
Description: as for outcome 4
Time Frame: 7 days after the M-TEL intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Interactive Multimedia Module | Power Point Show Module
Number analyzed (Participants) | 30 | 30
units on a scale | 1.0 [0.4 to 2.0] | 0.9 [0.3 to 1.9]

ADVERSE EVENTS:
Time Frame: We collected adverse event data 7 days after intervention.
Description: Because no previous adverse event of e-learning had been reported, we collected possible adverse event data using an anonymous qualitative feedback questionnaire.
Arm/Group | Interactive Multimedia Module | Power Point Show Module
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT02971735/Prot_SAP_000.pdf